CLINICAL TRIAL: NCT00928187
Title: Multicentric, Non-inferiority, Randomized, Non-blinded Phase 3 Trial Comparing Virological Response at 48 Weeks of 3 Antiretroviral Treatment Regimens in HIV-1-infected Patients With Treatment Failure After 1st Line Antiretroviral Therapy (Cameroon, Burkina Faso, Senegal)
Brief Title: Evaluation of Three Strategies of Second-line Antiretroviral Treatment in Africa (Dakar - Bobo-Dioulasso - Yaoundé)
Acronym: 2LADY
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Collaborators: Gilead Sciences (Industry); Janssen Pharmaceutica (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ANRS12169 2LADY
Record Dates: First submitted 2009-06-23; First posted 2009-06-25 (Estimated); Results first posted 2016-11-08 (Estimated); Last update posted 2017-02-27 (Actual); Status verified 2017-01

CONDITIONS: HIV; HIV Infections
Keywords: HIV; Second line treatment; WHO recommendations; Africa; Treatment strategies; treatment experienced
MeSH Terms: conditions — HIV Infections | interventions — Emtricitabine; Tenofovir; Lopinavir; abacavir; Didanosine; Ritonavir; Darunavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm A (Active Comparator): emtricitabine/tenofovir + lopinavir/ritonavir (WHO recommended second line)
  Interventions: Drug: emtricitabine/tenofovir + lopinavir/ritonavir (WHO recommended second line)
- Arm B (Active Comparator): abacavir + didanosine + lopinavir/ritonavir (WHO recommended second line)
  Interventions: Drug: abacavir + didanosine + lopinavir/ritonavir (WHO recommended second line)
- Arm C (Active Comparator): emtricitabine/tenofovir + darunavir + ritonavir (Second line strategy under evaluation)
  Interventions: Drug: emtricitabine/tenofovir + darunavir + ritonavir (Second line strategy under evaluation)

INTERVENTIONS:
Drug: emtricitabine/tenofovir + lopinavir/ritonavir (WHO recommended second line) — Emtricitabine 200 mg/tenofovir 300 mg 1 tablet/day with food + Lopinavir 200 mg/Ritonavir 50 mg 2 tablets in the morning and 2 tablets in the evening
  Arms: Arm A
Drug: abacavir + didanosine + lopinavir/ritonavir (WHO recommended second line) — Didanosine 1 entero-coated capsule/day in fasting conditions (dosage 250 mg if weight < 60 kg, 400 mg if weight > 60 kg) + abacavir 300 mg 1 tablet in the morning and in the evening + Lopinavir 200 mg/Ritonavir 50 mg 2 tablets morning and evening
  Arms: Arm B
Drug: emtricitabine/tenofovir + darunavir + ritonavir (Second line strategy under evaluation) — Emtricitabine 200 mg/tenofovir 300 mg 1 tablet/day with food + darunavir 400 mg 2 tablets + ritonavir 100 mg 1 capsule, in a single dose with food
  Arms: Arm C

SUMMARY:
Since the first line antiretroviral (ARV) treatment is now largely accessible in the Sub-Saharian Africa countries, documentation of virological failure, drug resistance patterns and second line treatment evaluation are still to be consolidated in settings where viral load monitoring is not available and non-B HIV subtype is predominant.

This trial aims at evaluating the efficacy and tolerance of 3 different second line treatment strategies: two recommended by WHO combine two non-nucleoside reverse transcriptase inhibitor associated with a ritonavir boosted protease inhibitor (emtricitabine-tenofovir-lopinavir/ritonavir and abacavir-didanosine-lopinavir/ritonavir); the third strategy combines emtricitabine-tenofovir-darunavir/ritonavir and is not yet evaluated in Sub-Saharian Africa. Darunavir has a potentially superior antiviral efficacy, a better tolerance and its single daily administration may facilitate treatment adherence.

ELIGIBILITY:
Inclusion Criteria:

* Patient over the age of 18 years at pre-inclusion and monitored under outpatient conditions
* Documented HIV-1 infection regardless of clinical stage and CD4 lymphocyte count
* Patient with treatment failure after first-line antiretroviral treatment with a combination including a non-nucleoside reverse transcriptase inhibitor and two nucleoside reverse transcriptase inhibitors, failure being defined as 2 measurements (at 1 month interval) of plasma HIV RNA levels > 1000 copies/ml after at least 6 months of uninterrupted treatment
* Adherence (> 80%) to first- line antiretroviral treatment (questionnaire) at pre inclusion
* Patient agrees not to take any concomitant medication during the trial without informing the investigator
* Informed consent signed no later than D-15
* For women in childbearing age: negative pregnancy test at inclusion, with no plan of pregnancy in the coming 12 months and agreeing to use mechanical contraception (with or without hormonal contraception) during the study

Exclusion Criteria:

* Infection with HIV-2 or HIV-1 groups O or N or HIV1+2
* Deficiency of the patient, making it difficult, if not impossible, for him/her to take part in the trial or understand the information provided to him/her
* Participation in any other clinical trial
* Presence of an uncontrolled, ongoing opportunistic infection or of any severe or progressive disease
* First-line treatment with a protease inhibitor, abacavir, tenofovir or ddI
* Ongoing treatment with rifampicin
* Severe hepatic insufficiency (TP < 50%)
* ALAT > 3 x ULN
* Creatinine clearance calculated by Cockcroft formula < 50 ml/min
* Hb ≤ 8 g/dl
* Platelets < 50,000 cells/mm3
* Neutrophiles < 500 cells/ mm3
* Use of drugs prohibited in the context of this trial (drugs contraindicated by the SCP of the trial drugs) - in the event of tuberculosis or malaria during the trial, a list of authorized medicines and, if necessary, a dose adjustment of the antiretroviral medication will be provided
* Pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 454 (Actual)
Dates: Start 2009-11; Primary Completion 2013-09 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sinata Koulla Shiro, PhD, Principal Investigator — Infectious diseases department, Central Hospital, Yaounde, Cameroon; Papa Salif Sow, PhD, Principal Investigator — Infectious Diseases Department, Fann Hospital, Dakar, Senegal; Adrien Sawadogo, MD, Principal Investigator — Day Hospital, CHU Sanou Souro, Bobo Dioulasso, Burkina Faso
Locations (3):
- Day Hospital, CHU Sanou Souro, Bobo-Dioulasso, Burkina Faso
- Day Hospital, Central Hospital, Yaoundé, Cameroon
- Clinical Research and Training Center, Fann Hospital, Dakar, Senegal

REFERENCES:
- [Derived] Boyer S, Nishimwe ML, Sagaon-Teyssier L, March L, Koulla-Shiro S, Bousmah MQ, Toby R, Mpoudi-Etame MP, Ngom Gueye NF, Sawadogo A, Kouanfack C, Ciaffi L, Spire B, Delaporte E; 2-Lady Group. Cost-Effectiveness of Three Alternative Boosted Protease Inhibitor-Based Second-Line Regimens in HIV-Infected Patients in West and Central Africa. Pharmacoecon Open. 2020 Mar;4(1):45-60. doi: 10.1007/s41669-019-0157-9. PMID 31273686

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment in three study sites (Yaoundé, Dakar and Bobo Dioulasso) in HIV day care clinics from January 2010 to September 2012.
Pre-assignment Details: 584 patients assessed for eligibility, 130 excluded primary (13.9%) because control viral load decreased below 1000 copies/mL after adherence support.
Period: Overall Study
Arm/Group | Arm A | Arm B | Arm C
Started | 152 | 147 | 155
Analysed | 152 | 145 | 154
Completed | 150 | 141 | 150
Not Completed | 2 | 6 | 5
Not completed — Death | 1 | 2 | 3
Not completed — Lost to Follow-up | 1 | 2 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 1
Not completed — Protocol Violation | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A | Arm B | Arm C | Total
Number analyzed (Participants) | 152 | 145 | 154 | 451
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 38 [34 to 45] | 38 [33 to 47] | 36 [32 to 45] | 38 [32 to 46]
Gender [Count of Participants; unit: Participants]
  Female | 113 | 105 | 106 | 324
  Male | 39 | 40 | 48 | 127
Region of Enrollment [Number; unit: participants]
  Cameroon | 101 | 99 | 102 | 302
  Burkina Faso | 30 | 28 | 32 | 90
  Senegal | 21 | 18 | 20 | 59
HIV RNA Viral Load [Median (Inter-Quartile Range); unit: log10 (copies/ml)] | 4.4 [4.0 to 5.0] | 4.6 [4.1 to 5.1] | 4.5 [4.0 to 5.1] | 4.5 [4.0 to 5.1]
Resistance to the three first-line drugs [Number; unit: participants] | 84 | 77 | 88 | 249
CD4 cells count [Median (Inter-Quartile Range); unit: cells/mm3] | 199 [92 to 318] | 195 [100 to 288] | 153 [81 to 261] | 183 [87 to 290]

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Plasma HIV RNA < 50 Copies/mL
Time Frame: 48 weeks
Population: ITT
Measure: Number; unit: participants
Arm/Group | Arm A | Arm B | Arm C
Number analyzed (Participants) | 152 | 145 | 154
participants | 105 | 92 | 97
Statistical Analysis 1: Comparison: Arm A vs Arm B; Test type: Non-Inferiority or Equivalence — Hypothesizing 80% efficacy at the 50 copies/mL Viral Load (VL) threshold in the control group at W48, we calculated a required sample size of 150 participants per group to show non-inferiority of ABC/ddI and DRV groups compared with control group in ITT analysis, with a non-inferiority margin of 15%, a power of 90% and a two-sided α of 5%; differences in proportions = 5.6, 95% CI 2-sided [-5.1 to 16.4]
Statistical Analysis 2: Comparison: Arm A vs Arm C; Test type: Non-Inferiority or Equivalence — Hypothesizing 80% efficacy at the 50 copies/mL VL threshold in the control group at W48, we calculated a required sample size of 150 participants per group to show non-inferiority of ABC/ddI and DRV groups compared with control group in ITT analysis, with a non-inferiority margin of 15%, a power of 90% and a two-sided α of 5%; difference in proportions = 6.1, 95% CI 2-sided [-4.5 to 16.7]

2. Secondary Outcome: Number of Patients With WHO Stage 3 and 4 HIV Related Events
Description: patients having a diagnosis of HIV related event classified as stage 3 or 4
Time Frame: between baseline and 48 weeks
Population: ITT
Measure: Number; unit: participants
Arm/Group | Arm A | Arm B | Arm C
Number analyzed (Participants) | 152 | 145 | 154
participants | 17 | 23 | 30

3. Secondary Outcome: Patients With Plasma HIV RNA < 200 Copies/ml
Description: number of patients with plasma HIV RNA below 200 copies/ml
Time Frame: 48 weeks
Population: ITT
Measure: Number; unit: participants
Arm/Group | Arm A | Arm B | Arm C
Number analyzed (Participants) | 152 | 145 | 154
participants | 130 | 118 | 127

4. Secondary Outcome: Gain in CD4 Cells Between Baseline and W48
Description: median gain in circulating CD4 cells between baseline and W48
Time Frame: between baseline and 48 weeks
Population: ITT with data available
Measure: Median (Inter-Quartile Range); unit: cell/mm3
Arm/Group | Arm A | Arm B | Arm C
Number analyzed (Participants) | 150 | 140 | 149
cell/mm3 | 133 [82 to 220] | 136 [78 to 206] | 115 [58 to 187]

5. Secondary Outcome: Number of Patients Discontinuing Study Treatment
Description: number of patients discounting treatment because of adverse events
Time Frame: between baseline and W48
Population: ITT
Measure: Number; unit: participants
Arm/Group | Arm A | Arm B | Arm C
Number analyzed (Participants) | 152 | 145 | 154
participants | 0 | 4 | 1

6. Secondary Outcome: Tolerance: Gastrointestinal Complains
Description: Gastrointestinal complaints (grade 1 to 4) between baseline and W48.
Time Frame: between baseline and 48 weeks
Population: ITT
Measure: Number; unit: participants
Arm/Group | Arm A | Arm B | Arm C
Number analyzed (Participants) | 152 | 145 | 154
participants | 50 | 48 | 26
Statistical Analysis 1: Comparison: Arm A vs Arm B vs Arm C; Test type: Superiority or Other; p = 0.001, Chi-squared

7. Secondary Outcome: Tolerance: Neuropathies (Grade 1 to 4)
Description: any symptom of peripheral neuropathy
Time Frame: between baseline and W48
Population: ITT
Measure: Number; unit: participants
Arm/Group | Arm A | Arm B | Arm C
Number analyzed (Participants) | 152 | 145 | 154
participants | 5 | 11 | 8
Statistical Analysis 1: Comparison: Arm A vs Arm B vs Arm C; Test type: Superiority or Other; p = 0.26, Chi-squared

8. Secondary Outcome: Tolerance: Equal or Superior to a 25% Reduction in eGFR (Glomerular Filtration Rate)
Description: evaluation of estimated glomerular filtration rate and number of participant with a decrease equal or superior to 25% of the baseline value
Time Frame: between baseline and W48
Population: ITT
Measure: Number; unit: participants
Arm/Group | Arm A | Arm B | Arm C
Number analyzed (Participants) | 152 | 145 | 154
participants | 28 | 14 | 19
Statistical Analysis 1: Comparison: Arm A vs Arm B vs Arm C; Test type: Superiority or Other; p = 0.13, Chi-squared

9. Secondary Outcome: Adherence
Description: number of patients in different categories of adherence as measured by questionnaire
Time Frame: between baseline and W48
Population: patients with data available
Measure: Number; unit: participants
Arm/Group | Arm A | Arm B | Arm C
Number analyzed (Participants) | 150 | 140 | 159
participants
  Always above 95% | 50 | 54 | 67
  At least once 80-95% | 89 | 72 | 78
  At least once < 80% | 11 | 14 | 4

10. Secondary Outcome: Number of Patients With Resistance Mutations
Description: number of patients with resistance mutations after second line treatment failure (HIV RNA> 1000 copies/ml)
Time Frame: between W12 and W48
Population: patients who failed second line (2 HIV RNA measure above 1000 copies/ml)
Measure: Number; unit: participants
Arm/Group | Arm A | Arm B | Arm C
Number analyzed (Participants) | 2 | 2 | 1
participants | 0 | 0 | 0

11. Secondary Outcome: Development of Metabolic Syndrome
Description: number of patients developing metabolic syndrome over a period of 48 weeks
Time Frame: from baseline to week 48
Population: population with data available
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B | Arm C
Number analyzed (Participants) | 143 | 132 | 144
Participants | 12 | 21 | 9

12. Secondary Outcome: Number of Patients With HIV Plasma Viral Load < 50 Copies/ml
Description: Snapshot of patients with HIV viral load less then 50 copies/ml at week 24
Time Frame: Week 24
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B | Arm C
Number analyzed (Participants) | 152 | 145 | 154
Participants | 90 | 81 | 97

13. Secondary Outcome: Number of Patients With HIV Plasma Viral Load < 200 Copies/ml
Description: number of patients having a plasma viral load below 200 copies/ml at week 24
Time Frame: Week 24
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B | Arm C
Number analyzed (Participants) | 152 | 145 | 154
Participants | 127 | 117 | 129

ADVERSE EVENTS:
Time Frame: 48 Weeks
Description: SAE grade 3, grade 4 and hospitalisation
Arm/Group | Arm A | Arm B | Arm C
Serious Adverse Events (participants affected / at risk) | 13/152 | 22/145 | 19/154
Other Adverse Events (participants affected / at risk) | 131/152 | 122/145 | 118/154
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (N=152) | Arm B (N=145) | Arm C (N=154)
Intracranial injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Acute posthemorrhagic anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Other anaemias (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 3 (3)
Pulmonary embolism (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Unspecified diabetes mellitus (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Other functional intestinal disorders (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Other noninfective gastroenteritis and colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal and pelvic pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Abnormal findings on diagnostic imaging of lung (General disorders) | 0 (0) | 1 (1) | 0 (0)
Abnormal serum enzyme levels (General disorders) | 1 (1) | 0 (0) | 0 (0)
Abnormalities of breathing (General disorders) | 0 (0) | 0 (0) | 1 (1)
Cough (General disorders) | 0 (0) | 1 (2) | 1 (1)
Elevated blood glucose level (General disorders) | 0 (0) | 1 (1) | 0 (0)
Fever of other and unknown origin (General disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (General disorders) | 0 (0) | 1 (1) | 1 (1)
Malaise and fatigue (General disorders) | 2 (2) | 1 (1) | 1 (1)
Pain in throat and chest (General disorders) | 0 (0) | 2 (2) | 1 (1)
Symptoms and signs concerning food and fluid intake (General disorders) | 0 (0) | 0 (0) | 1 (1)
Unattended death (General disorders) | 1 (1) | 2 (2) | 1 (1)
Infectious gastroenteritis and colitis, unspecified (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Other septicaemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Respiratory tuberculosis, bacteriologically and histologically confirmed (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Respiratory tuberculosis, not confirmed bacteriologically or histologically (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Tuberculosis of other organs (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Unspecified malaria (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Medical observation and evaluation for suspected diseases and conditions (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Unspecified severe protein- calorie malnutrition (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Volume depletion (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Malignant neoplasm of liver and intrahepatic bile ducts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Other abnormal products of conception (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1)
Spontaneous abortion (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 2 (2) | 0 (0)
Acute renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Acute tubulo-interstitial nephritis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Other disorders of urinary system (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0)
Unspecified renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Excessive, frequent and irregular menstruation (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Salpingitis and oophoritis (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Bacterial pneumonia, not elsewhere classified (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Pneumonia in diseases classified elsewhere (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumonia, organism unspecified (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure, not elsewhere classified (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Cutaneous abscess, furuncle and carbuncle (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Lichen simplex chronicus and prurigo (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (N=152) | Arm B (N=145) | Arm C (N=154)
Agranulocytosis (Blood and lymphatic system disorders) | 12 (13) | 7 (8) | 7 (8)
Other functional intestinal disorders (Gastrointestinal disorders) | 16 (19) | 14 (18) | 5 (5)
Other noninfective gastroenteritis and colitis (Gastrointestinal disorders) | 14 (15) | 4 (4) | 1 (1)
Abdominal and pelvic pain (General disorders) | 9 (9) | 16 (18) | 8 (8)
Cough (General disorders) | 17 (19) | 11 (15) | 16 (21)
Fever of other and unknown origin (General disorders) | 9 (9) | 8 (9) | 4 (4)
Headache (General disorders) | 14 (16) | 14 (17) | 16 (19)
Malaise and fatigue (General disorders) | 11 (12) | 9 (9) | 7 (8)
Nausea and vomiting (General disorders) | 8 (8) | 13 (14) | 6 (6)
Pain, not elsewhere classified (General disorders) | 9 (10) | 5 (5) | 5 (6)
Symptoms and signs concerning food and fluid intake (General disorders) | 28 (37) | 24 (28) | 11 (11)
Candidiasis (Infections and infestations) | 5 (5) | 12 (18) | 13 (16)
Infectious gastroenteritis and colitis, unspecified (Infections and infestations) | 33 (37) | 22 (25) | 10 (14)
Unspecified malaria (Infections and infestations) | 17 (19) | 10 (13) | 9 (9)
Contraceptive management (Injury, poisoning and procedural complications) | 10 (11) | 5 (5) | 7 (10)
Pregnancy examination and test (Injury, poisoning and procedural complications) | 5 (5) | 8 (8) | 5 (7)
Dorsalgia (Musculoskeletal and connective tissue disorders) | 14 (14) | 4 (4) | 4 (4)
Other joint disorders, not elsewhere classified (Musculoskeletal and connective tissue disorders) | 6 (8) | 12 (12) | 7 (7)
Other polyneuropathies (Nervous system disorders) | 4 (4) | 10 (10) | 8 (8)
Other inflammation of vagina and vulva (Reproductive system and breast disorders) | 9 (9) | 8 (9) | 5 (5)
Acute bronchitis (Respiratory, thoracic and mediastinal disorders) | 19 (19) | 15 (16) | 11 (12)
Acute nasopharyngitis [common cold] (Respiratory, thoracic and mediastinal disorders) | 9 (12) | 7 (7) | 7 (7)
Influenza, virus not identified (Respiratory, thoracic and mediastinal disorders) | 20 (22) | 15 (18) | 16 (19)
Cutaneous abscess, furuncle and carbuncle (Skin and subcutaneous tissue disorders) | 12 (14) | 3 (4) | 5 (5)
Lichen simplex chronicus and prurigo (Skin and subcutaneous tissue disorders) | 12 (14) | 9 (10) | 14 (14)
Pruritus (Skin and subcutaneous tissue disorders) | 18 (19) | 24 (26) | 18 (22)

LIMITATIONS AND CAVEATS:
Limitations: open label design, random imbalance at baseline. Non-inferiority not shown, results influenced by the hypothesis of 80% viral success (50 copies/mL), not reached (69% in the control group). Therefore, the study power was reduced (80%).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No